CLINICAL TRIAL: NCT04459468
Title: Identify Proteomic Biomarkers for Outcome Prediction of Locoregional Treatments for Hepatocellular Carcinoma (HCC)
Brief Title: Identify Proteomic Biomarkers for Outcome Prediction of Locoregional Treatments for HCC
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Anil Pillai, ASSOC PROFESSOR - Radiology, University of Texas Southwestern Medical Center
Other Study IDs: STU-2019-1758
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ethiodized Oil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pre and Post-treatment procedure blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- HCC for Lipiodol TACE, denovo ablation, or Y90 radioembolization: These patients will receive standard of care Lipiodol TACE, denovo ablation, or Y90 radioembolization treatment. No research intervention is planned.
  Interventions: Drug: Lipiodol
- Healthy controls: Healthy controls from public database
- HCC patients: HCC patients will be used for biomarker validation.

INTERVENTIONS:
Drug: Lipiodol — Lipiodol TACE procedure
  Groups: HCC for Lipiodol TACE, denovo ablation, or Y90 radioembolization

SUMMARY:
This study will enroll patients with hepatocellular carcinoma being planned for TACE or other standard of care treatment (such as denovo ablation or Y90) and obtain blood samples pre and post treatment procedure for biomarker identification using bead based X-aptamer library. No intervention is planned.

DETAILED DESCRIPTION:
This is a prospective, non-blinded, multi-arm study. Patients at 18 - 70 years old with liver cancer will be enrolled.

The approach is to identify novel proteomic biomarkers for HCC patients treated with Lipiodol TACE, denovo ablation or Y90 using beads-based X-aptamer library, then validate and create a biomarker panel that can be used to predict the outcome of HCC post treatment.

Lipiodol TACE, denovo ablation, or Y90 will be done as standard of care and the only thing done as research will be blood draws pre and post-TACE.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent.
2. Male or female aged 18-70years.
3. Diagnosed with primary or metastatic liver cancer.
4. Scheduled to undergo Lipoidal TACE, denovo ablation, or Yttrium-90 (Y90) radioembolization as part of standard of care.

Exclusion Criteria:

Subjects who have received chemotherapy, radiation or surgery for HCC.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Predictive accuracy of Proteomic biomarker(s) measured with bead-based X-aptamer library for overall survival in hepatocellular carcinoma patients | 2 years
  X-aptamer identified biomarker to predictability for tumor response rate after treatment with Lipoidol TACE compared to standard of care biomarkers-AFP.

SECONDARY OUTCOMES:
Predictive accuracy of Proteomic biomarker(s) measured with bead-based X-aptamer library for Progression free survival in Hepatocellular carcinoma patients. | 2 years
  X-aptamer identified biomarker to predict overall survival after treatment with Lipoidol TACE .

CONTACTS AND LOCATIONS:
Overall Officials: Anil Pillai, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided